CLINICAL TRIAL: NCT02941120
Title: Retrospective Observational Study for Reconstruction of Localized, Full-thickness Cartilage Defects in the Knee Joint With In-situ Polymerizable and Chondrocyte Populated Biomaterial (NOVOCART® Inject)
Brief Title: Non-interventional Study With NOVOCART® Inject in the Reconstruction of the Knee Cartilage Defects
Acronym: RENOVO
Status: Completed | Type: Observational
Sponsor: Tetec AG (Industry)
Collaborators: Aesculap AG (Industry); Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1521
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-01

CONDITIONS: Cartilage Disease
Keywords: Cartilage defect; Knee; ACT (Autologous chondrocyte implantation); NOVOCART® Inject
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NOVOCART® Inject patients: Patients who where treated with NOVOCART® Inject autologous chondrocyte implantation in the knee joint.

SUMMARY:
Retrospective non-interventional study to evaluate safety and efficacy of NOVOCART® Inject in patients with full-thickness cartilage defects in the knee joint.

DETAILED DESCRIPTION:
Retrospective and multicenter non-interventional study to evaluate safety and efficacy of NOVOCART® Inject in patients with localized full-thickness cartilage defects in the knee joint.

Safety: Measuring the number of adverse drug reactions/serious adverse drug reactions since treatment and up to the present time.

Efficacy: Evaluate symptoms and functional status at the present time using IKDC 2000 (International Knee Documentation Committee) and KOOS (Knee injury osteoarthritis outcome score).

ELIGIBILITY:
Inclusion Criteria:

* male and female patients
* juvenile patients with closed epiphysial plate
* insulated full-thickness cartilage damage of the knee Joint, ICRS (International Cartilage Repair Society) grade 3-4
* defect size ≥ 2.5 and ≤ 10 cm2
* intact or reconstructed bony subchondral plate
* in the case of deep bony substance defects, additional bony reconstruction is needed

Exclusion Criteria:

* radiographic signs of osteoarthritis of Kellgren and Lawrence > 2
* joint stiffness
* arthrofibrosis
* malalignment in the knee (valgus- or varus deformity) > 3° (correction contemporary to the ACT)
* insufficient reconstructed ligaments (correction contemporary to the ACT)
* defective position patella (correction contemporary to the ACT)
* sled prosthesis implants or carbon pin
* inflammatory joint diseases (f.e. rheumatoid arthritis)
* corresponding cartilage defects ("kissing lesions")
* more than two independent cartilage defects in one knee
* primary cartilage reconstructive treatment in children and juvenile with open epiphysial plate
* diffuse chondromalacia
* congenital or gained deformity of patella

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Orthopaedic clinics
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Number of adverse drug reaction/serious adverse drug reaction | Up to 24 months
  Number of adverse drug reaction/serious adverse drug reaction as a measurement of safety

SECONDARY OUTCOMES:
Outcome of IKDC 2000 | Up to 24 months
  Outcome of the IKDC 2000 as measurements of symptoms and function
Outcome of KOOS | Up to 24 months
  Outcome of KOOS as measurements of symptoms and function

CONTACTS AND LOCATIONS:
Locations (7):
- Germany (7):
  - Hochtaunus-Kliniken gGmbH Krankenhaus Bad Homburg, Bad Homburg
  - Gelenk-Klinik Gundelfingen, Gundelfingen
  - Orthopädische Praxisklinik im Zentrum, Kelkheim
  - Orthopädische Klinik Markgröningen gGmbH, Markgröningen
  - Dr. med. Michael Moraldo, Dr. med. Sebastian Lauber, Münster
  - Nordwest-Krankenhaus Sanderbusch gGmbH, Sande
  - Muldentalkliniken GmbH Krankenhaus Wurzen, Wurzen

IPD SHARING:
Plan to Share IPD: Undecided